CLINICAL TRIAL: NCT00736866
Title: A Pragmatic Randomized Clinical Trial Evaluating the Effect of Acetylcysteine for Contrast-induced Nephropathy
Brief Title: The Acetylcysteine for Contrast-Induced Nephropathy Trial
Acronym: ACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Medley Pharmaceutical Industry SA (Unknown)
Responsible Party: Otavio Berwanger, Hospital do Coracao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IEP- HCor 001/08
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2008-08

CONDITIONS: Acute Kidney Failure
Keywords: acetylcysteine; contrast-induced nephropathy; angiography; angioplasty with or without Stent
MeSH Terms: conditions — Acute Kidney Injury | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetylcysteine (Experimental)
  Interventions: Drug: Acetylcysteine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylcysteine — Acetylcysteine: 1200 mg every 12 hours for a total of 4 doses. Treatment is to be started 12 hours before angiography, that is, two doses should be administered before it. When this is not achievable, at least one dose should be administered before angiography.
  Arms: Acetylcysteine
Drug: Placebo — Placebo of Acetylcysteine: every 12 hours PO, for a total of 4 doses. Treatment is to be started 12 hours before angiography, that is, two doses should be administered before it. When this is not achievable, at least one dose should be administered before angiography.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy of acetylcysteine compared to placebo for the contrast-induced nephropathy prevention, between 48 and 96 hours after procedures that use contrast.

Contrast-induced nephropathy is defined as an increase of 25% in serum creatinine before the procedure.

ELIGIBILITY:
Inclusion Criteria:

At least one of the following criteria:

* Aged more than 70 years-old
* Chronic renal failure (defined as serum creatinine higher than 1.5mg/dL within the last 3 months)
* Diabetes mellitus
* Congestive heart failure or ventricular disfunction (left ventricular ejection fraction less than 0.45)
* Shock or intra-aortic balloon pump use
* Urgency or emergency procedures

Exclusion Criteria:

* Pregnant women, breastfeeding or aged below 45 years-old and with no efficacious contraceptive methods.
* Patients in dialysis
* Previous inclusion in this trial
* Patient refusal to informed consent
* Pacientes com Infarto Agudo do Miocárdio com supradesnivelamento do segmento S-T nos quais não seja possível administrar o protocolo de hidratação pré e pós-procedimento.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Contrast-induced nephropathy incidence | between 48 and 96 hours after angiographic procedures

SECONDARY OUTCOMES:
Combined outcome of total mortality, dialysis indication or basal serum creatinine duplication | within 30 days
Combined outcome of total mortality or dialysis indication | within 30 days
The individual components of the combined outcome | within 30 dias

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Sousa, PhD, Principal Investigator — Hospital do Coracao
Locations (1):
- Hospital do Coração, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Berwanger O, Cavalcanti AB, Sousa AM, Buehler A, Castello-Junior HJ, Cantarelli MJ, Mangione JA, Bergo RR, Sao Thiago LE, Nunes PM, da Motta PA, Kodama A, Victor E, Carvalho VO, Sousa JE; Acetylcysteine for Contrast-Induced Nephropathy Trial Investigators. Acetylcysteine for the prevention of renal outcomes in patients with diabetes mellitus undergoing coronary and peripheral vascular angiography: a substudy of the acetylcysteine for contrast-induced nephropathy trial. Circ Cardiovasc Interv. 2013 Apr;6(2):139-45. doi: 10.1161/CIRCINTERVENTIONS.112.000149. Epub 2013 Apr 9. PMID 23572490
- [Derived] ACT Investigators. Acetylcysteine for prevention of renal outcomes in patients undergoing coronary and peripheral vascular angiography: main results from the randomized Acetylcysteine for Contrast-induced nephropathy Trial (ACT). Circulation. 2011 Sep 13;124(11):1250-9. doi: 10.1161/CIRCULATIONAHA.111.038943. Epub 2011 Aug 22. PMID 21859972
- [Derived] ACT Trial Investigators. Rationale, design, and baseline characteristics of the Acetylcystein for Contrast-Induced nephropaThy (ACT) Trial: a pragmatic randomized controlled trial to evaluate the efficacy of acetylcysteine for the prevention of contrast-induced nephropathy. Trials. 2009 Jun 4;10:38. doi: 10.1186/1745-6215-10-38. PMID 19497091